CLINICAL TRIAL: NCT00062543
Title: Hepatic Artery Infusion of CD34+ Cells, Isolated by the Isolex 300i Device, in Stem Cell Transplant Recipients With Hepatic Failure Due to Veno-occlusive Disease
Brief Title: Hepatic Artery Infusion of CD34+ Cells
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-167
Record Dates: First submitted 2003-06-09; First posted 2003-06-12 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Stem Cell Transplantation; Liver Diseases
Keywords: Severe hepatic dysfunction post stem cell transplantation; Stem Cell Transplantation; Hepatic Artery Infusion; Liver Diseases; CD34+ Cells; SCT
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hepatic Artery Infusion (Experimental): Donor-derived CD34+ cells administered in a total volume of 100ml via hepatic artery over 10 minutes. Cells given as a dose escalation study. First cohort of 3 patients receive 1 * 106 CD34+ cells/kg. Next 3 patients receive 2.5 * 106 CD34+cells/kg. Next 3 patients receive 5 * 106 CD34+ cells/kg. Less than 1 * 105 T cells/kg administered.
  Interventions: Procedure: Hepatic artery infusion of CD34+ cells; Device: Cobe Spectra

INTERVENTIONS:
Procedure: Hepatic artery infusion of CD34+ cells — Donor's cells infused directly into liver through a groin catheter (hepatic artery).
Device: Cobe Spectra — Mononuclear cells (MNC) collected by continuous-flow centrifugation using a blood cell separator (Cobe Spectra).
  Other Names: blood cell separator

SUMMARY:
The primary objective is to determine whether donor stem cells administered via hepatic artery infusion can produce liver cells in patients with severe hepatic dysfunction post stem cell transplantation (SCT) and the safety of this procedure. The secondary objective is to improve liver function and improve survival.

DETAILED DESCRIPTION:
Participants in this study have received stem cell transplantation. As a result of this procedure, participants have developed severe liver dysfunction. Researchers have recently discovered that cells circulating in the blood and bone marrow are capable of forming liver cells. Before taking part in this study, women able to have children must have a negative blood pregnancy test.

Participants in this study will have donor's cells infused directly into their liver through a catheter that will be inserted through the groin. This will be done after liver disease has been diagnosed by liver biopsy. The catheter will stay in the groin for no more than 3 days. During that time, participants will be exposed to repeated x-ray exams to ensure that the catheter stays in place.

During the time that the catheter is in place, the infusion will be repeated as long as donor's cells are available. Participants will receive different drugs by vein to decrease the risk of transfusion reaction. After completing donor cell infusion, the catheter will be removed.

After participants are released from the hospital, they will have periodic evaluation of liver size. About 1 teaspoon of blood will be drawn for standard blood tests to evaluate liver function. Around Days 28 and 90, participants will have liver biopsy.

This is an investigational study. A total of 10 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

* SCT recipients with severe hepatic dysfunction (bilirubin equal to or greater than 5mg/dl) and histologically documented VOD.
* The original stem cell donor must be sex-mismatched, willing and able to donate G-CSF-mobilized peripheral blood stem cells.
* The patient must have complete donor chimerism.

Exclusion Criteria:

* Patients who do not have at least 5 x 10^6 donor CD34+ cells/kg available for infusion.
* Patients with graft versus host disease (GVHD).
* Patients in whom hepatic artery infusion cannot be performed because of anatomical or technical reasons.
* Patients with active hepatitis B or C.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Learn if donor's cells can produce liver cells when injected directly into the liver and whether this procedure will improve liver function and survival. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Estrov, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org